CLINICAL TRIAL: NCT06408662
Title: Remote Delivery of a Mindfulness-based Intervention for Tics
Acronym: MBIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Bowdoin College (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00413599; R01AT012455 (NIH)
Record Dates: First submitted 2024-05-06; First posted 2024-05-10 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Tourette Syndrome; Tourette's Disorder; Chronic Motor Tic Disorder; Chronic Vocal Tic Disorder; Persistent Motor Tic Disorder; Persistent Vocal Tic Disorder; Persistent Tic Disorder; Tic Disorders
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: This project is a randomized controlled trial (RCT) that will compare the efficacy of a mindfulness-based intervention for tics (MBIT) to psychoeducation with relaxation and supportive therapy (PRST) in 150 adults with TS. The study interventions will be delivered in a group format and provided remotely using a secure telehealth services platform. The study assessments will be completed using a secure telehealth services platform and online electronic data capture systems. An independent evaluator (IE) masked to treatment condition will administer all assessments during the treatment and follow-up periods.
Who Masked: Outcomes Assessor
Masking Description: The independent evaluator (IE) will conduct study related assessments during the treatment and follow-up periods, and will be masked to treatment condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mindfulness-based intervention for tics (MBIT) (Experimental): This is an 8-week mindfulness-based group intervention delivered via telehealth. It consists of mindfulness and meditative practice, didactics, inquiry, discussion and weekly therapeutic exercises and assignments (i.e., homework).
  Interventions: Other: mindfulness-based intervention for tics (MBIT)
- psychoeducation with relaxation and supportive therapy (PRST) (Active Comparator): This is an 8-week educational and supportive therapy group intervention delivered via telehealth. It consists of psychoeducation, relaxation, discussion, and weekly therapeutic exercises and assignments (i.e., homework).
  Interventions: Other: psychoeducation with relaxation and supportive therapy (PRST)

INTERVENTIONS:
Other: mindfulness-based intervention for tics (MBIT) — Psychological intervention that focuses on cultivating awareness of urges to tic and developing a different relationship to those urges through meditation and other mindfulness practice
  Arms: mindfulness-based intervention for tics (MBIT)
Other: psychoeducation with relaxation and supportive therapy (PRST) — Psychological Intervention that focuses on learning more about tics, practicing a range of strategies for coping with tics (e.g., relaxation, effective communication), and discussing challenges commonly experienced by individuals with tics.
  Arms: psychoeducation with relaxation and supportive therapy (PRST)

SUMMARY:
This research study is being done to compare a mindfulness-based intervention for tics (MBIT) to psychoeducation with relaxation and supportive therapy (PRST) for individuals with Tourette's syndrome or Persistent Tic Disorders (collectively TS). It is the investigator's hope that this information cam be used to improve current treatments for individuals with TS.

DETAILED DESCRIPTION:
Tourette's syndrome and other persistent tic disorders (collectively, TS) is a condition that onsets in childhood and affects ~1% of the population. Alongside motor and vocal tics, patients with TS experience distressing somatosensory sensations (i.e., premonitory urges) and co-occurring mental health conditions such as anxiety disorders, depressive disorders, obsessive-compulsive disorder (OCD), and ADHD. Tics and comorbid symptoms cause individuals with TS significant distress and impairment across life domains (e.g., physical, social, academic, occupational, emotional, and familial). Two evidence-based treatments exist for TS: behavior therapy and pharmacotherapy. Behavior therapy [often referred to as habit reversal training (HRT) or the comprehensive behavioral intervention for tics (CBIT)] is an evidence-based treatment that has been shown to reduce the severity of tic symptoms, and has a low risk for adverse effects. Although behavior therapy is recognized as a first-line intervention for TS, less than 40% of adults with TS respond to this evidence-based treatment. Additionally, current behavioral interventions are often inaccessible for adults with TS. While pharmacotherapy for tic management (e.g., antipsychotic medications) has been shown to be effective, these treatments can have adverse side effects with detrimental health consequences. Thus, there is a critical need for new treatments for adults with TS that are efficacious for reducing tic severity, beneficial for co-occurring conditions, and have few adverse health effects. Mindfulness-based interventions have proven beneficial for adults with a wide range of neuropsychiatric conditions. Based on the investigator's prior work, the investigators believe that a mindfulness-based intervention for tics (MBIT) is beneficial for adults with TS.

This project is a randomized controlled trial (RCT) that will compare the efficacy of a mindfulness-based intervention for tics (MBIT) to psychoeducation with relaxation and supportive therapy (PRST) in 150 adults with TS. All interventions and assessments will be delivered remotely using secure telehealth services platforms and online electronic data capture systems. An independent evaluator (IE) masked to treatment condition will administer all assessments during the treatment and follow-up periods. The investigators will test the mechanisms by which MBIT reduces tic severity, and examine the efficacy of MBIT relative to PRST for common co-occurring psychiatric symptoms and quality of life impairments-towards "treating the whole person". Finally, the investigators will explore the sustained therapeutic improvement from MBIT over a 6-month follow-up period focusing on tic severity, tic-related impairment, co-occurring psychiatric symptoms, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. be ≥18 years of age;
2. meet diagnostic criteria for a primary or co-primary diagnosis of Tourette Syndrome or a Persistent Motor or Vocal Tic Disorder on a structured clinical interview;
3. have moderate or greater tic severity as evidenced by a YGTSS Total Tic Score of >14 (when motor and vocal tics are present) or >10 (when only motor or vocal tics are present);
4. be medication free and/or on a stable dose of psychiatric medication 8 weeks prior to study participation;
5. be not engaged in psychotherapy for non-TS conditions and/or be on a stable course of therapy for 6 months prior to study participation
6. be fluent in English;
7. have access to a smart phone and/or tablet.

Exclusion Criteria:

1. a current diagnosis of substance use disorder, psychosis, mania or another condition that requires another form of care;
2. severe current suicidal/homicidal ideation and/or self-injury requiring medical intervention;
3. concurrent psychotherapy for TS;
4. prior extensive experience with mindfulness and/or meditation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Yale Global Tic Severity Scale (YGTSS) Total Tic Severity Score | Screen, Baseline (Week 0), Mid-treatment (Week 5), Post-treatment (Week 9), 1-month follow-up (Week 13), 3-month follow-up (Week 22), and 6-month follow-up (Week 35)
  The YGTSS is a clinician-administered measure of tic symptom severity (0-50) and impairment (0-50). Greater scores are reflective of greater severity and/or impairment.

SECONDARY OUTCOMES:
Clinical Global Impressions Scales of Severity and Improvement (CGI-S & CGI-I) | Screen, Baseline (Week 0), Mid-treatment (Week 5), Post-treatment (Week 9), 1-month follow-up (Week 13), 3-month follow-up (Week 22), and 6-month follow-up (Week 35)
  In order for a participant to be considered a treatment responder, he or she must receive a score of 1 (not ill or very much improved) or 2 (borderline mentally ill or much improved).
Adult Tic Questionnaire (ATQ) | Screen, Baseline (Week 0), Mid-treatment (Week 5), Post-treatment (Week 9), 1-month follow-up (Week 13), 3-month follow-up (Week 22), and 6-month follow-up (Week 35)
  Higher ATQ scores reflect a worse outcome. For each tic present in the past week, its severity score is the sum of its frequency score (0-4, 4 worst, occurring "almost all the time during the day") and its intensity score (0-4, 4 worst). The ATQ severity score is the sum of the severity score for each of up to 27 tics present in the past week. The minimum possible severity score on the ATQ is 0, indicating that no tics were present in the past week. The maximum possible severity score on the ATQ indicates is 216, indicating that a tic of each of the 27 types listed was present in the past week, each with an item severity score of 8 = 4 + 4.
Yale-Brown Obsessive Compulsive Scale-II | Baseline (Week 0), Mid-treatment (Week 5), Post-treatment (Week 9), 1-month follow-up (Week 13), 3-month follow-up (Week 22), and 6-month follow-up (Week 35)
  A clinician-administered measure of OCD severity that has shown good psychometric properties. The total score ranges from 0 to 50, with greater total score reflective of greater severity.
Attention-Deficit Hyperactivity Rating Scale (ADHD-RS) | Baseline (Week 0), Mid-treatment (Week 5), Post-treatment (Week 9), 1-month follow-up (Week 13), 3-month follow-up (Week 22), and 6-month follow-up (Week 35)
  A self-report measure of ADHD severity that has shown good psychometric properties in TS studies. The total score ranges from 0 to 72, with greater scores indicating greater ADHD severity.
Patient Health Questionnaire-9 (PHQ-9) | Baseline (Week 0), Mid-treatment (Week 5), Post-treatment (Week 9), 1-month follow-up (Week 13), 3-month follow-up (Week 22), and 6-month follow-up (Week 35)
  A self-report measure of depressive symptom severity (range: 0-27), with greater total score reflecting greater depressive severity.
Premonitory Urge to Tic Scale (PUTS) | Baseline (Week 0), Mid-treatment (Week 5), Post-treatment (Week 9), 1-month follow-up (Week 13), 3-month follow-up (Week 22), and 6-month follow-up (Week 35)
  A self-report measure of premonitory urges (range: 0-36), with a greater total score reflective of greater premonitory urges.
Five Facet Mindfulness Questionnaire (FFMQ) | Baseline (Week 0), Mid-treatment (Week 5), Post-treatment (Week 9), 1-month follow-up (Week 13), 3-month follow-up (Week 22), and 6-month follow-up (Week 35)
  Each item is rated on a 1 to 5 scale with 1=never or very rarely true and 5=very often or always true; responses are summed and then divided by 39 (the number of items). Higher scores on the FFMQ reflects a higher level of mindfulness (a better outcome).
Client Satisfaction Questionnaire | Post-treatment (Week 9)
  An 8-item self-report measure assessing client's satisfaction with treatment services. The total score ranges from 8 to 32. Greater total score corresponds with greater satisfaction with services
Self Compassion Scale | Baseline (Week 0), Mid-treatment (Week 5), Post-treatment (Week 9), 1-month follow-up (Week 13), 3-month follow-up (Week 22), and 6-month follow-up (Week 35)
  Measure ranges from 26 to 130, with higher scores indicating higher levels of self-compassion
Affective Reactivity Index | Baseline (Week 0), Mid-treatment (Week 5), Post-treatment (Week 9), 1-month follow-up (Week 13), 3-month follow-up (Week 22), and 6-month follow-up (Week 35)
  A 6-item scale of affective reactivity that ranges from 0-12, with higher scores reflective of greater affective reactivity.
Brief Irritability Test | Baseline (Week 0), Mid-treatment (Week 5), Post-treatment (Week 9), 1-month follow-up (Week 13), 3-month follow-up (Week 22), and 6-month follow-up (Week 35)
  A five-item self-report measure of irritability that ranges from 5 to 30, with greater scores reflective of greater irritability.

OTHER OUTCOMES:
Individualized Premonitory Urge to Tic Scale (I-PUTS) | Screen, Baseline (Week 0), Mid-treatment (Week 5), Post-treatment (Week 9), 1-month follow-up (Week 13), 3-month follow-up (Week 22), and 6-month follow-up (Week 35)
  The I-PUTS is a clinician-administered scale that parallels the YGTSS symptom checklist. The clinician assesses each tic that is present in the past week for premonitory urges. The urges are rated on the dimensions of frequency (1-4) and intensity (1-4), with the frequency and intensity summed to create a total premonitory urge severity score
Depression Anxiety and Stress Scale (DASS) | Screen, Baseline (Week 0), Mid-treatment (Week 5), Post-treatment (Week 9), 1-month follow-up (Week 13), 3-month follow-up (Week 22), and 6-month follow-up (Week 35)
  The Depression Anxiety and Stress Scale (DASS) is a self-report measure of depression, anxiety, and stress. The 21-items are rated on a scale from 0 to 2, with a total score ranging from 0 to 42. Greater scores are reflective of worse symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph F McGuire, PhD, Principal Investigator — Johns Hopkins University; Hannah Reese, PhD, Principal Investigator — Bowdoin College
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No